CLINICAL TRIAL: NCT03496246
Title: Vitamin D Status in Inflammatory Bowel Disease
Acronym: vdsinibd
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohammed ragab, resident doctor at internal medicine department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2929mroam
Record Dates: First submitted 2018-04-01; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Vitamin D Deficiency; Inflammatory Bowel Diseases
MeSH Terms: conditions — Vitamin D Deficiency; Inflammatory Bowel Diseases | interventions — Blood Cell Count; Blood Sedimentation

STUDY DESIGN:
Intervention Model Description: It is a Clinical trial with three arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): patients with vitamin D deficiency are investigated for serum total 25 hydroxycholecalciferol 25(OH) vitamin D,complete blood count (CBC),serum calcium level ,serum phosphurus level,erythrocyte sedimentation rate (ESR),C-reactive protein (CRP),serum creatinine ,serum albumin level,seum alanine aminotransferase and serum potassium level.
  Interventions: Diagnostic Test: serum total 25 hydroxycholecalciferol 25(OH) vitamin D; Diagnostic Test: complete blood count (CBC); Diagnostic Test: serum calcium level; Diagnostic Test: erythrocyte sedimentation rate (ESR); Diagnostic Test: C-reactive protein (CRP); Diagnostic Test: serum creatinine; Diagnostic Test: serum albumin level; Diagnostic Test: seum alanine aminotransferase; Diagnostic Test: serum potassium level; Diagnostic Test: serum phosphurus level
- Group B (Active Comparator): patients with vitamin D insufficiency are investigated for serum total 25 hydroxycholecalciferol 25(OH) vitamin D,complete blood count (CBC),serum calcium level ,serum phosphurus level,erythrocyte sedimentation rate (ESR),C-reactive protein (CRP),serum creatinine ,serum albumin level,seum alanine aminotransferase and serum potassium level.
  Interventions: Diagnostic Test: serum total 25 hydroxycholecalciferol 25(OH) vitamin D; Diagnostic Test: complete blood count (CBC); Diagnostic Test: serum calcium level; Diagnostic Test: erythrocyte sedimentation rate (ESR); Diagnostic Test: C-reactive protein (CRP); Diagnostic Test: serum creatinine; Diagnostic Test: serum albumin level; Diagnostic Test: seum alanine aminotransferase; Diagnostic Test: serum potassium level; Diagnostic Test: serum phosphurus level
- Group C (Active Comparator): patients with normal vitamin D level normal are investigated for serum total 25 hydroxycholecalciferol 25(OH) vitamin D,complete blood count (CBC),serum calcium level ,serum phosphurus level,erythrocyte sedimentation rate (ESR),C-reactive protein (CRP),serum creatinine ,serum albumin level,seum alanine aminotransferase and serum potassium level.
  Interventions: Diagnostic Test: serum total 25 hydroxycholecalciferol 25(OH) vitamin D; Diagnostic Test: complete blood count (CBC); Diagnostic Test: serum calcium level; Diagnostic Test: erythrocyte sedimentation rate (ESR); Diagnostic Test: C-reactive protein (CRP); Diagnostic Test: serum creatinine; Diagnostic Test: serum albumin level; Diagnostic Test: seum alanine aminotransferase; Diagnostic Test: serum potassium level; Diagnostic Test: serum phosphurus level

INTERVENTIONS:
Diagnostic Test: serum total 25 hydroxycholecalciferol 25(OH) vitamin D — Quantitative measurement of serum total 25(OH) vitamin D by ELISA. Fasting (6-8 hours), venous blood samples(10ml) are collected from participants in the morning and after centrifugation, the serum are preserved in the deep freezer at -20 c. Serum levels will be determined by using commercially available kits.
Diagnostic Test: complete blood count (CBC) — for measurement of hemoglobin level and white blood cell count percent of neutrophils ,lymphocytes and esoinphils
Diagnostic Test: serum calcium level — measurement of total calcium level after correction with albumin level as it is closely related to vitamin d with its effects on its level
Diagnostic Test: erythrocyte sedimentation rate (ESR) — it is an indicator of activity in inflammatory bowel disease
Diagnostic Test: C-reactive protein (CRP) — it is an indicator for increased possibility of infections
Diagnostic Test: serum creatinine — for assessment of renal function
Diagnostic Test: serum albumin level — for possibility of malabsorbtion in patients with inflammatory bowel disease
Diagnostic Test: seum alanine aminotransferase — for assessment of liver function
Diagnostic Test: serum potassium level — indicator for hypokalemia increased in patients with diarrhea as result of inflammatory bowel disease
Diagnostic Test: serum phosphurus level — measurement of phosphurus level as it is closely related to vitamin d with its effects on its level

SUMMARY:
Inflammatory bowel disease (IBD), comprising crohn's disease (CD) and ulcerative colitis (UC), is a a chronic, relapsing-remitting systemic disease. Vitamin D is a secosteroid hormone that possesses immunomodulatory properties and has been demonstrated to potentially influence inflammatory bowel disease (IBD) pathogenesis and activity.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), comprising crohn's disease (CD) and ulcerative colitis (UC), is a a chronic, relapsing-remitting systemic disease and it is increasing sharply with rapidly increasing proportion in developing countries., and the common medications are not effective for most patients.The key underlying pathogenic mechanisms for both diseases is a dysregulated host immune response to commensal intestinal flora in genetically susceptible individuals.Vitamin D is a fat-soluble vitamin, a secosteroid hormone whose active form, calcitriol or 1,25-dihydroxyvitaminD3 (1,25(OH)2D3) plays important roles in immune regulation, particularly involving the innate immune system, cell differentiation and intercellular adhesion, promotes the production of anti-microbial peptides, including β-defensins and cathelicidins, the shift towards Th2 immune responses, and regulates autophagy and epithelial barrier integrity.The relationship between vitamin D deficiency and IBD is bidirectional that vit D with its immunomodulatory effects influence IBD pathogenesis and activity and IBD itself can lead to vitamin D deficiency.Vitamin D deficiency has associated with increased IBD activity scores, lower quality-of-life, an increased risk of IBD-related surgery and increased hospitalizations.[4]. Vitamin D downregulate powerful proinflammatory cytokines, such as TNF, which enhance the durability of anti-TNF therapy in IBD and its deficency has been found to be associated with earlier cessation of anti-TNFα therapy( loss of response to biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with Inflammatory Bowel Disease (either ulcerative colitis or crohns disease ) patients diagnosed through clinical evaluation ,laboratory ,colonoscopic and histopathological studies.

Exclusion Criteria:

* patients known to have malignancy, or metabolic disease associated with vitamin D and calcium abnormalities e.g. hyperparathyroidism and history of vitamin D supplementations.
* patients with known biliary disease, chronic liver and kidney diseases.
* Patients with a mal-absorption syndrome other than IBD.
* Pregnant or lactating patients.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
vitamin D deficency in Inflammatory Bowel Disease | one day
  serum total 25(OH) vitamin D is measured in patients with Inflammatory Bowel Disease (either ulcerative colitis or crohns disease) by Quantitative measurement by ELISA with Fasting (6-8 hours), venous blood samples will be collected from participants in the morning. Serum 25(OH)D levels of less than 20 ng/mL indicate vitamin D deficiency.
vitamin D insufficiency in Inflammatory Bowel Disease | one day
  by Quantitative measurement of serum total 25(OH) vitamin D by ELISA with Fasting (6-8 hours), venous blood samples will be collected from participants in the morning. Serum 25(OH)D levels between 21 and 29 ng/mL indicate vitamin D insufficiency.

SECONDARY OUTCOMES:
the severity of Inflammatory Bowel Disease with its relation to vitamin D level the severity is detected by a composite clinical and biomarker index called the Seo index | one day
  severity of Inflammatory Bowel Disease is detected by a composite clinical and biomarker index that combines the clinical symptoms including fever, bleeding and stool frequency with biomarkers including C-reactive protein (CRP), erythrocyte sedimentation rate(ESR),complete blood count (CBC), serum electrolytes.
  we will investigate the relation between vitamin D deficiency and severity of Inflammatory Bowel Disease

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Ragab Osman, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burisch J, Munkholm P. Inflammatory bowel disease epidemiology. Curr Opin Gastroenterol. 2013 Jul;29(4):357-62. doi: 10.1097/MOG.0b013e32836229fb. PMID 23695429
- [Background] Ananthakrishnan AN. Environmental risk factors for inflammatory bowel diseases: a review. Dig Dis Sci. 2015 Feb;60(2):290-8. doi: 10.1007/s10620-014-3350-9. Epub 2014 Sep 10. PMID 25204669
- [Background] Abraham BP, Prasad P, Malaty HM. Vitamin D deficiency and corticosteroid use are risk factors for low bone mineral density in inflammatory bowel disease patients. Dig Dis Sci. 2014 Aug;59(8):1878-84. doi: 10.1007/s10620-014-3102-x. Epub 2014 Mar 12. PMID 24619280
- [Background] Ananthakrishnan AN, Cagan A, Gainer VS, Cai T, Cheng SC, Savova G, Chen P, Szolovits P, Xia Z, De Jager PL, Shaw SY, Churchill S, Karlson EW, Kohane I, Plenge RM, Murphy SN, Liao KP. Normalization of plasma 25-hydroxy vitamin D is associated with reduced risk of surgery in Crohn's disease. Inflamm Bowel Dis. 2013 Aug;19(9):1921-7. doi: 10.1097/MIB.0b013e3182902ad9. PMID 23751398
- [Background] Zator ZA, Cantu SM, Konijeti GG, Nguyen DD, Sauk J, Yajnik V, Ananthakrishnan AN. Pretreatment 25-hydroxyvitamin D levels and durability of anti-tumor necrosis factor-alpha therapy in inflammatory bowel diseases. JPEN J Parenter Enteral Nutr. 2014 Mar-Apr;38(3):385-91. doi: 10.1177/0148607113504002. Epub 2013 Oct 2. PMID 24088707
- [Background] Holick MF. The vitamin D deficiency pandemic: Approaches for diagnosis, treatment and prevention. Rev Endocr Metab Disord. 2017 Jun;18(2):153-165. doi: 10.1007/s11154-017-9424-1. PMID 28516265
- [Background] Rosen CJ. Clinical practice. Vitamin D insufficiency. N Engl J Med. 2011 Jan 20;364(3):248-54. doi: 10.1056/NEJMcp1009570. No abstract available. PMID 21247315
- [Background] Farraye FA, Nimitphong H, Stucchi A, Dendrinos K, Boulanger AB, Vijjeswarapu A, Tanennbaum A, Biancuzzo R, Chen TC, Holick MF. Use of a novel vitamin D bioavailability test demonstrates that vitamin D absorption is decreased in patients with quiescent Crohn's disease. Inflamm Bowel Dis. 2011 Oct;17(10):2116-21. doi: 10.1002/ibd.21595. Epub 2011 Jan 6. PMID 21910173
- [Background] Ulitsky A, Ananthakrishnan AN, Naik A, Skaros S, Zadvornova Y, Binion DG, Issa M. Vitamin D deficiency in patients with inflammatory bowel disease: association with disease activity and quality of life. JPEN J Parenter Enteral Nutr. 2011 May;35(3):308-16. doi: 10.1177/0148607110381267. PMID 21527593
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Bernstein CN, Leslie WD. Review article: Osteoporosis and inflammatory bowel disease. Aliment Pharmacol Ther. 2004 May 1;19(9):941-52. doi: 10.1111/j.1365-2036.2004.01876.x. PMID 15113361
- [Background] Shih DQ, Targan SR. Immunopathogenesis of inflammatory bowel disease. World J Gastroenterol. 2008 Jan 21;14(3):390-400. doi: 10.3748/wjg.14.390. PMID 18200661